CLINICAL TRIAL: NCT02041416
Title: Delivering the Geriatric Assessment Tool to Older Adults With Cancer Using Computer Survey Methodologies: Testing Feasibility, Reliability, and Validity of Research Electronic Data Capture (REDCap) and Support Screen (Touchscreen) Technologies
Brief Title: Technology to Assess Vulnerable Older Adults With Cancer and Their Caregivers
Status: Active, not recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 13103; R21AG041489 (NIH)
Record Dates: First submitted 2014-01-03; First posted 2014-01-22 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Solid Tumor; Hematologic Malignancy
Keywords: Geriatric assessment; REDCap; touchscreen; age 65
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Group 1: REDCap and paper pencil
- Group 2: REDCap twice
- Group 3: Support Screen and paper pencil
- Group 4: Support Screen twice

SUMMARY:
The goal of this study is to determine the feasibility, reliability, and validity of administering the Geriatric Assessment Tool using these two different computer based survey platforms, REDCap and Support Screen. The development of a computer based Geriatric Assessment Tool has the potential to improve research and clinical practice by providing an efficient user friendly means to collect and analyze data for geriatric oncology patients.

DETAILED DESCRIPTION:
Sixty percent of all cancer diagnoses and 70% of all cancer mortality occurs in patients age 65 and older. Patients older than age 65 years have an 11-fold increased cancer incidence and a 16-fold increase in cancer mortality in comparison to those younger than 65 years. The population at risk is growing rapidly: the number of adults age 65 years and older is expected to double in the next 30 years. In order to adequately care for this growing population of older adults, oncologists need an assessment tool that provides information regarding an older individual's "functional age" rather than just "chronological age." The Geriatric Assessment Tool developed by Hurria and colleagues has been found to help identify those older adults who are more vulnerable to complications from cancer treatment.

The Geriatric Assessment Tool takes into account well validated measures of functional status, co-morbid medical conditions, cognitive function, psychological state, nutritional status, social activity, and social support. Pilot data demonstrates the feasibility of this assessment which can be completed in less than 30 minutes; however, this assessment is completed by pencil and paper, and therefore requires an interviewer to deliver, score, and summarize the assessment results. The development of a computer based Geriatric Assessment Tool would have practical importance for both research and clinical practice. It could potentially allow more efficient data collection and analysis in the research setting. In turn it would potentially influence clinical decision making by medical oncologists given its ability to predict chemotherapy related toxicity among geriatric oncology patients across all tumor types.

Two electronic platforms have been developed for the Geriatric Assessment Tool:

1. Research Electronic Data Capture (REDCap) is a secure website designed by Vanderbilt University that is used by 48 countries, and 511 institutions around the world including research centers that comprise the Cancer and Aging Research Group. REDCap is a web-based application that allows researchers to build and manage online surveys and databases. It also provides a central web-based forum where data can be processed uniformly and efficiently. Administering the Geriatric Assessment Tool through REDCap would potentially improve data collection and analysis for elderly cancer patients across multiple research centers.
2. Support Screen is a program developed by researchers and information technology specialists at City of Hope utilizing touchscreen technology to deliver patient surveys. The touchscreen platform has been used in previous studies as a means of assessing the needs of cancer patients. Support Screen is an attractive technology given it is user friendly for patients and has the unique capability of transferring information from the touchscreen device directly into the City of Hope medical record system in a secure, HIPPA-compliant manner, thereby providing clinicians and researchers real time access to survey information. A pilot study looking at the feasibility of delivering the Geriatric Assessment to elderly cancer patients using Support Screen has been performed at City of Hope with promising results, but the reliability and validity of this modality have yet to be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients age ≥65 with any performance status
* Diagnosis of cancer (solid tumor or hematologic malignancy)
* Able to provide informed consent

Exclusion Criteria:

• Non-English speaking because some components of the geriatric assessment tool have not yet been validated in other languages.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Using a prospective longitudinal study design, 100 patients will be recruited for this study from the outpatient medical oncology and hematology practice at City of Hope Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-05-15 (Actual); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Patient's ability to complete the assessment | 2 years
  Measured by responses to questionnaire. To be determined by the patient's ability to complete the assessment without assistance, the length of time it takes to complete the assessment, the mean number of missing items and patient satisfaction.
Item correlation between different assessment platforms | 2 years
  Measured by responses to questionnaire. Test for item correlations greater than 0.7 versus a null hypothesis of correlation.
Positive correlations between different measures of functional status | 2 years
  Internal consistency using Cronbach's alpha and Pearson's correlation.

SECONDARY OUTCOMES:
Questionnaire- percentage of patients who did not enter the study and the reason for declining participation | 2 years
  Determine if there are different demographic characteristics among those who decline versus participate. Patients who decline participation in the study will be asked for permission to capture the following demographic information: 1) age, 2) gender, 3) race, 4) ethnicity, and 5) reason for declining enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States